CLINICAL TRIAL: NCT00389766
Title: International Phase II Studies of I-mIBG in Combination With Topotecan and Peripheral Blood Stem Cell Rescue for (A) Primary Resistant High Risk Neuroblastoma and (B) Relapsed Stage 4 Neuroblastoma
Brief Title: High-Dose Iodine I 131 Metaiodobenzylguanidine, Topotecan, and Peripheral Stem Cell Transplant in Treating Young Patients With Relapsed Stage 4 Neuroblastoma or Primary Resistant High-Risk Neuroblastoma
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Withdrawn because protocol has been discontinued. It was never opened.
Sponsor: Children's Cancer and Leukaemia Group (Other)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CCLG-NB-2006-08; CDR0000508611 (Registry Identifier: PDQ (Physician Data Query)); EU-20644; EUDRACT-2005-002089-13
Record Dates: First submitted 2006-10-18; First posted 2006-10-19 (Estimated); Last update posted 2013-07-10 (Estimated); Status verified 2007-06

CONDITIONS: Neuroblastoma
Keywords: localized unresectable neuroblastoma; recurrent neuroblastoma; regional neuroblastoma; localized resectable neuroblastoma; disseminated neuroblastoma
MeSH Terms: conditions — Neuroblastoma | interventions — 3-Iodobenzylguanidine; Topotecan; Drug Therapy; Peripheral Blood Stem Cell Transplantation; Whole-Body Irradiation

INTERVENTIONS:
Drug: iodine I 131 metaiodobenzylguanidine
Drug: topotecan hydrochloride
Procedure: chemotherapy
Procedure: peripheral blood stem cell transplantation
Procedure: radioisotope therapy
Procedure: radionuclide imaging
Procedure: radiosensitization
Procedure: total-body irradiation

SUMMARY:
RATIONALE: Radioisotope therapy, such as iodine I 131 metaiodobenzylguanidine (MIBG), releases radiation that kills tumor cells. Drugs used in chemotherapy, such as topotecan, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Topotecan may also make tumor cells more sensitive to iodine I 131 MIBG. A peripheral stem cell transplant may be able to replace blood-forming cells that were destroyed by iodine I 131 MIBG and topotecan. This may allow more iodine I 131 MIBG and topotecan to be given so that more tumor cells are killed.

PURPOSE: This phase II trial is studying how well giving high-dose iodine I 131 MIBG together with topotecan and peripheral stem cell transplant works in treating young patients with relapsed stage 4 neuroblastoma or primary resistant high-risk neuroblastoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine response (partial and complete response at metastatic sites) in children with relapsed stage 4 neuroblastoma or primary resistant high-risk neuroblastoma treated with high-dose iodine I 131 metaiodobenzylguanidine, topotecan hydrochloride, and peripheral blood stem cell transplantation.
* Determine the proportion of patients who, as a result of this treatment, are able to progress to potentially curative surgery and further systemic treatment.
* Correlate tumor dosimetry (to determine whether the tumor absorbed the radiation dose) with response in patients treated with this regimen.
* Determine the time to tumor progression.

OUTLINE: This is an open-label, multicenter study. Patients are stratified according to disease type (relapsed stage 4 vs primary resistant high-risk neuroblastoma).

Patients receive topotecan hydrochloride IV over 30 minutes on days 1-5 and 15-19 and high-dose iodine I 131 metaiodobenzylguanidine (^131I-MIBG) IV over 30 minutes on days 1 and 15. Patients receive autologous CD 34+ peripheral blood stem cells when ^131I-MIBG dosimetry levels reach an acceptable low on days 25-29.

Total whole-body absorbed dose is measured periodically after the first ^131I-MIBG dose is administered and periodically thereafter.

After completion of study treatment, patients are followed periodically for up to 10 years.

PROJECTED ACCRUAL: A total of 67 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Confirmed diagnosis of neuroblastoma meeting the 1 of the following criteria:

  * Primary resistant high-risk disease meeting the following criteria:

    * International neuroblastoma staging system (INSS) stage 4, or stage 2 or 3 with myelocytomatosis viral-related oncogene (MycN) amplification
    * Failed to achieve satisfactory remission with induction chemotherapy, defined as one of the following:

      * Less than 50% reduction or > 3 positive sites on iodine I 131 metaiodobenzylguanidine (^131I-MIBG) scintigraphy
      * Persistent cytomorphological positive disease in bone marrow aspirates or trephine biopsies
      * Progressive disease necessitating a change of treatment
  * Relapsed stage 4 disease meeting the following criteria:

    * High-risk neuroblastoma (INSS stage 4, or stage 2 or 3 with MycN amplification)
    * Relapsed after intensive treatment including high-dose chemotherapy and hematopoietic progenitor cell support

      * Patients may be entered at the time of relapse, or at any point subsequently after other treatments
* ^131I-MIBG-positive disease on diagnostic scintigraphy
* Peripheral blood stem cell harvest ≥ 300,000/mm³ CD 34+ cells
* Enrolled in or has been treated on protocol SIOP-NB-2009 or a similar protocol

PATIENT CHARACTERISTICS:

* Glomerular filtration rate ≥ 50 mL/min
* Considered fit enough to undergo proposed study treatment

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2008-07; Primary Completion 2008-07 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients who respond to treatment (partial response and complete response at metastatic sites) as measured by metaiodobenzylguanidine scintigraphy and positron emission tomography and CT imaging
Proportion of patients who are able to progress to potentially curative treatment with surgery and further systemic treatment
Correlation of tumor dosimetry with response
Time to tumor progression

CONTACTS AND LOCATIONS:
Overall Officials: Mark N. Gaze, MD, Study Chair — University College London Hospitals